CLINICAL TRIAL: NCT03676595
Title: Effects of Interactive Video Game-Based Exercise on Balance in Diabetic Patients With Peripheral Neuropathy
Brief Title: Video Game Balance Training for Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201308020
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Neuropathy Peripheral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received interactive video game-based exercise training for the first 6 weeks, with no exercise in the subsequent 6 weeks. The exercise program consisted of 30-minute sessions 3 times per week for 6 weeks. Outcomes were measured at weeks 0, 6, and 12.
  Interventions: Other: interactive video game-based exercise; Other: no exercise
- Group B (Experimental): Group B had no exercise in the first 6 weeks and then underwent interactive video game-based exercise training in the subsequent 6 weeks. The exercise program consisted of 30-minute sessions 3 times per week for 6 weeks. Outcomes were measured at weeks 0, 6, and 12.
  Interventions: Other: interactive video game-based exercise; Other: no exercise

INTERVENTIONS:
Other: interactive video game-based exercise — Twenty-four patients were randomly assigned to two groups (12 participants per group). Group A received interactive video game-based exercise training for the first 6 weeks, with no exercise in the subsequent 6 weeks. Group B had no exercise for the first 6 weeks and then underwent interactive video game-based exercise training in the subsequent 6 weeks.
Other: no exercise — Twenty-four patients were randomly assigned to two groups (12 participants per group). Group A received interactive video game-based exercise training for the first 6 weeks, with no exercise in the subsequent 6 weeks. Group B had no exercise for the first 6 weeks and then underwent interactive video game-based exercise training in the subsequent 6 weeks.

SUMMARY:
This study evaluated the effects of interactive video game-based exercise (IVGB) on balance in diabetic patients with peripheral neuropathy. Twenty-four patients were randomly assigned to two groups (12 participants per group). Group A received IVGB training for the first 6 weeks, with no exercise in the subsequent 6 weeks. Group B had no exercise for the first 6 weeks and then underwent IVGB training in the subsequent 6 weeks. Both subjective and objective measures were used to determine whether IVGB exercise improves balance function.

DETAILED DESCRIPTION:
Participants in Group A received IVGB intervention for the first 6 weeks (intervention phase), with no exercise in the subsequent 6 weeks (control phase), whereas participants in Group B received no IVGB intervention in the first 6 weeks (control phase), followed by 6 weeks of IVGB intervention (intervention phase). The IVGB intervention protocol consisted of 30-minute training sessions comprising four tasks designed to focus on lower limb strength, balance, and coordination training. Balance assessments consisted of both subjective and objective measures, including the Modified Falls Efficacy Scale (MFES), Time Up and Go (TUG) test, Berg Balance Scale (BBS), and Unipedal Stance Test (UST). For all participants, these tests were conducted at weeks 0, 6, and 12 of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* medical diagnoses of diabetes under regular medication control and diabetic peripheral neuropathy confirmed using an electrodiagnostic test
* independent community ambulatory individuals
* intact cognition (Mini-Mental State Examination score of >24).

Exclusion Criteria:

* other neurological diseases such as dementia, Parkinson's disease, spinal cord injury, or stroke;
* severe visual impairment, musculoskeletal disorders, unhealed plantar ulceration, lower limb amputation, poor cardiopulmonary function, or other diseases affecting walking ability or any other disease due to which individuals were unable to walk without assistance
* any other condition associated with a high risk of falling.
* Inability to follow simple instructions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change of Berg Balance Scale (BBS) score | 15 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  It consists of 14 functional tasks of varying difficulty, including sitting, standing, changing posture, transfers, reaching forward, retrieving objects, turning, tandem stance, and one-leg stance. It is a valid tool used in both clinical practice and research to evaluate the efficacy of intervention and provide a quantitative description of balance function. The ability to perform each a task is scored on a scale of 0-4, ranging from inability to independently perform the task to successfully completing it, respectively. The maximum possible score for the 14 functional tasks is 56.

SECONDARY OUTCOMES:
Change of Time Up and Go (TUG) test time | 5 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  Participants stand up from a 46-cm-high armchair with back support, walk straight for 3 m, turn around, walk back to the chair, and sit down as quickly and safely as possible. The timing starts when the investigator says "go" and stops when the participant sits back down on the chair. In our study, each participant had three chances to complete the TUG test in each session, and the best result was recorded for each participant.
Change of Modified Falls Efficacy Scale (MFES) scores | 10 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  MFES is a 14-item questionnaire related to daily indoor and outdoor physical activities. It is a 10-point visual analog scale of confidence level in completing a particular activity (item) without falling, rated from 0 to 10, where 0 denotes not confident or sure at all, and 10 denotes completely confident or sure. The total score for the 14 items ranges from 0 to 140.
Change of Unipedal Stance Test (UST) time | 5 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  Participants raised one leg to the ankle level or higher without touching the other leg or using any assistance and then stood on that leg for as long as possible barefoot and with eyes open. The observer measured the length of time for which participants maintained balance; that is, until they were no longer able to keep the leg raised at or above the ankle level or when both legs touched the ground. The observer stopped counting at 45 seconds, recording this as the time for any participant who maintained balance for a longer time. Each participant performed the test three times for both right and left legs, with the best result for each leg recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, Principal Investigator — Taipei Medical University Hospital

IPD SHARING:
Plan to Share IPD: Undecided